CLINICAL TRIAL: NCT03717714
Title: A Randomized, Double-blind, Active Controlled, 12-week Follow-up, Pilot Study to Evaluate the Safety and Efficacy of Polycan in Combination With Glucosamine for Treatment of Knee Osteoarthritis
Brief Title: Polycan in Combination With Glucosamine for Treatment of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vietstar Biomedical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Polycan-VN01
Record Dates: First submitted 2018-10-20; First posted 2018-10-24 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Glucosamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Glucosamine 1500mg (Active Comparator): Glucosamine 1500 mg per day for 12 weeks
  Interventions: Dietary Supplement: Glucosamine 1500 mg
- Polycan & Glucosamine 750mg (Experimental): Polycan 50 mg + Glucosamine 750 mg per day for 12 weeks
  Interventions: Dietary Supplement: Polycan 50mg + Glucosamine 750 mg
- Polycan & Glucosamine 1500mg (Experimental): Polycan 50 mg + Glucosamine 1500 mg per day
  Interventions: Dietary Supplement: Polycan 50mg + Glucosamine 1500 mg

INTERVENTIONS:
Dietary Supplement: Glucosamine 1500 mg — Patients in this group take 3 capsules, each capsule contains Placebo 16.7mg and Glucosamine 500 mg, once a day for 12 weeks
  Arms: Glucosamine 1500mg
Dietary Supplement: Polycan 50mg + Glucosamine 750 mg — Patients in this group take 3 capsules, each capsule contains Polycan 16.7mg and Glucosamine 250 mg, once a day for 12 weeks
  Arms: Polycan & Glucosamine 750mg
Dietary Supplement: Polycan 50mg + Glucosamine 1500 mg — Patients in this group take 3 capsules, each capsule contains Polycan 16.7mg and Glucosamine 500 mg, once a day for 12 weeks
  Arms: Polycan & Glucosamine 1500mg

SUMMARY:
The objectives of this study is to examine the Safety and Eﬃcacy of black yeast beta-glucan produced from Aureobusidium pulluluns SM-2001 (Polycan), in combination with glucosamine in reducing knee osteoarthritis (OA) associated symptoms. This study is a double-blind, randomized, active-controlled trial conducted with 100 OA patients, aged 35-80 years using a formulated product

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of knee osteoarthritis (OA)
* OA ranging from grade 1 to grade 3 by Kellgren and Lawrence system
* Agree to participate into the study

Exclusion Criteria:

* OA ranging from grade 4 by Kellgren and Lawrence system
* Allergic or contradicted with oral NSAIDs (Meloxicam)
* Pregnant and breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) changes at 12 weeks in the three groups | Baseline to Week 12
  The WOMAC consists of 24 items divided into 3 subscales:
  Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing Stiffness (2 items): after first waking and later in the day Physical Function (17 items): stair use, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy household duties, light household duties.
  Total WOMAC score ranges from 0 to 96 with higher scores indicate worse pain, stiffness, and functional limitations

SECONDARY OUTCOMES:
Number of dose of rescue medication (Meloxicam 7.5mg) used in the three groups. | Through study completion, an average of 12 weeks
  Rescue medication (Meloxicam 7.5mg) used by patients for 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- 198 Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided